CLINICAL TRIAL: NCT05686174
Title: Investigation on Safety and Efficacy of Soybean Fermented Extract (MBS217) in Treating Patients With Non-alcoholic Fatty Liver Disease: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study in National Taiwan University Hospital
Brief Title: Investigation on Safety and Efficacy of Soybean Fermented Extract (MBS217) in Treating Patients With NAFLD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202108126RIPB
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBS-217 (Active Comparator): 4 ml MBS-217 twice a day for 16 weeks
  Interventions: Dietary Supplement: MBS217
- Placebo (Placebo Comparator): 4 ml MBS-217 placebo twice a day for 16 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MBS217 — Soybean Fermented Extract (MBS217)
  Arms: MBS-217
Dietary Supplement: Placebo — Without active ingredient
  Arms: Placebo

SUMMARY:
Investigators aimed to investigate the efficacy and safety of fermented soybean extract (MBS-217) in treating participants with Non-alcoholic fatty liver disease (NAFLD) in this study.

DETAILED DESCRIPTION:
Background: NAFLD is one of the most prevalent chronic liver diseases in Taiwan. NAFLD can progress to fibrosis, cirrhosis, and even liver cancer. Based on the current trend in epidemiology, fatty liver disease is forecasted to be the leading cause of liver transplantation by 2030. Since NAFLD imposes a significant medical burden and there is no approved medication for NAFLD, developing an effective therapy for improving NAFLD is undoubtedly an unmet need. Diet and gut microbiota play pivotal roles in NAFLD progress. The composition of the gut microbiota and gut barrier function is affected by dietary factors, which cause pathophysiological impacts on the liver through the immune and metabolic communications between gut and liver, which is coined as the "gut-liver axis." Therefore, intervention with dietary products from probiotics and prebiotics may be an opportunity to develop effective therapy against NAFLD. In fact, current evidence has shown that fermented soybean products can modulate hepatic lipid metabolism and possess potential prebiotic activities. Also, our preliminary data have shown that MBS217 supplementation has the effects of modulating gut microbiota and regulating the hepatic inflammatory-related immune response in both nonalcoholic steatohepatitis (NASH) mice and healthy adult subjects. Objective: Investigators aimed to investigate the efficacy and safety of MBS217 in treating participants with NAFLD in this study. The changes in other metabolic parameters, gut microbiome, metabolomics, and gut permeability will also be investigated. Methods: Using a block randomization with a block size of 2 in a 1:1 ratio, 30 eligible adult subjects aged 20-70 years diagnosed with NAFLD will be randomized to receive one of the following regimens. This study plans to enroll 30 eligible adult subjects aged 20-70 years diagnosed with NAFLD. Enrolled subjects will be randomly assigned to receive 4 mL of either MBS217 or placebo (1:1) treatment for 16 weeks and then followed for 8 weeks, with assessment for NAFLD-related parameters, gut microbiome, metabolomics, and gut permeability. Outcome analysis: The primary outcome is the improvement of hepatic steatosis, fibrosis, stiffness, and FIB-4 evaluated by FibroScan or MRI. The secondary outcomes are the frequency of adverse events, the overall NAFLD-related parameters, gut microbiota, metabolomics, and gut permeability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 20 and 70 years old.
* Serum ALT of the subject is between 40-200 U/L.
* The subject is diagnosed as NAFLD through FibroScan (CAP > 220 db/m).
* BMI of the subject is between 18.5-40 kg/m2.
* The subject is able to provide written informed consent by himself/herself and agrees to comply with all protocol requirements.
* The subject agrees to comply with the following two requirements:

comply with all follow-up visit requirements according to the trial protocol. comply with all requirement regarding fecal samples collection, storage and delivery according to the trial protocol.

* If the subject is reproductive women, she should agree to take more than two ways of contraceptive methods.

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject has received any antibiotic (excluding topical agents), antifungals or antivirals within 30 days prior to visit 1.
* The subject has received any steroids (excluding topical agents), immunosuppressant or anti-inflammation drugs within 14 days prior to visit 1.
* The subject has received probiotics or prebiotics 14 days prior to visit 1.
* The subject has received medication affecting evaluating indicators, including hepatitis and lipid metabolism related compounds, but excluding the following medicines: Statins, Fibrates, Silymarin, N-Acetyl Cystein, Thiazolidinediones, Metformin, Fibrate, Cholestyramine, Ezetimibe, Orlistat, SGLT2i and GLP1-RAs.
* The subject has a clinically significant, currently active or underlying diarrhea (loose stools more than three times in 24 hours) of infectious etiologies.
* The subject who has been diagnosed a severe/injury hepatic disease, acute/chronic viral hepatitis B, acute/chronic viral hepatitis C, human immunodeficiency virus infection, disease affecting liver function, active inflammatory bowel disease, gastric ulcer, chronic kidney disease, kidney function repairmen, chronic gut inflammatory disease, coronary artery disease with arterial stent surgery in half year, cancer, autoimmune disease, fasting glucose≥ 300 mg/dl, HbA1c>9%, or serum triglyceride≥ 500 mg/dl.
* The subject currently is participating in studies involving other investigational drugs, medical devices, functional foods, or cosmetic within 30 days prior to visit 1.
* The subject has participated in body weight control plan within 60 days prior to visit 1.
* The subject has an alcohol abuse problem.
* The subject has been aboard for 10 days within 60 days prior to visit 1, or plans to go aboard during this study.
* The subject has soybean allergy.
* The subject is vegetarian or special diet.
* The subject is considered by the investigator as not suitable for the trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota | baseline to 8th, 12th, 16th and 24th weeks
  evaluated by fecal 16S rRNA gene sequencing
Improvement of intrahepatic fibrosis | baseline to 16th and 24th weeks
  evaluated by FibroScan
Changes in hepatic steatosis composition | baseline to 16th week
  evaluated by MRI-PDFF and MRI-MRS

SECONDARY OUTCOMES:
Changes in FIB-4 | baseline to 12th, 16th and 24th weeks
  Fibrosis-4 (FIB-4) Index
Changes in gut permeability | baseline to 16th week
  evaluated by lactulose/mannitol ratio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang SC, Su HJ, Kao JH, Tseng TC, Yang HC, Su TH, Chen PJ, Liu CJ. Clinical and Histologic Features of Patients with Biopsy-Proven Metabolic Dysfunction-Associated Fatty Liver Disease. Gut Liver. 2021 May 15;15(3):451-458. doi: 10.5009/gnl20218. PMID 33431715